CLINICAL TRIAL: NCT06140758
Title: Evaluation of the Anticaries Efficacy of Various Dentifrice Formulations Using an In-situ Model
Brief Title: Evaluation of the Anticaries Efficacy of Dentifrice Formulations Using an In-situ Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022085
Record Dates: First submitted 2023-11-14; First posted 2023-11-20 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Caries
MeSH Terms: interventions — fluorophosphate; Dentifrices; Tin Fluorides

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Oral-B 1450 ppm Fluoride (1.16% sodium monofluorophosphate) Dentifrice (Active Comparator)
  Interventions: Drug: Oral-B 1450 ppm Fluoride (1.16% sodium monofluorophosphate) Dentifrice
- Colgate 1450 ppm Fluoride (1.16% sodium monofluorophosphate)Dentifrice (Active Comparator)
  Interventions: Drug: Colgate 1450 ppm Fluoride (1.16% sodium monofluorophosphate)Dentifrice
- Toms of Maine 0 ppm Fluoride Dentifrice (Sham Comparator)
  Interventions: Drug: Toms of Maine 0 ppm Fluoride Dentifrice
- Colgate 1450 ppm Fluoride (1.1% sodium monofluorophosphate) Dentifrice (Active Comparator)
  Interventions: Drug: Colgate 1450 ppm Fluoride (1.1% sodium monofluorophosphate) Dentifrice
- 1500 ppm MFP/CaCO3 1.16% sodium monofluorophosphate) Dentifrice (Active Comparator)
  Interventions: Drug: 1500 ppm MFP/CaCO3 1.16% sodium monofluorophosphate) Dentifrice
- 1100 ppm (0.454% Stannous fluoride) Dentifrice (Active Comparator)
  Interventions: Drug: 1100 ppm (0.454% Stannous fluoride) Dentifrice

INTERVENTIONS:
Drug: Oral-B 1450 ppm Fluoride (1.16% sodium monofluorophosphate) Dentifrice — Each subject will use this product during one of the six treatment periods in the crossover study design.
  Arms: Oral-B 1450 ppm Fluoride (1.16% sodium monofluorophosphate) Dentifrice
Drug: Colgate 1450 ppm Fluoride (1.16% sodium monofluorophosphate)Dentifrice — Each subject will use this product during one of the six treatment periods in the crossover study design.
  Arms: Colgate 1450 ppm Fluoride (1.16% sodium monofluorophosphate)Dentifrice
Drug: Toms of Maine 0 ppm Fluoride Dentifrice — Each subject will use this product during one of the six treatment periods in the crossover study design.
  Arms: Toms of Maine 0 ppm Fluoride Dentifrice
Drug: Colgate 1450 ppm Fluoride (1.1% sodium monofluorophosphate) Dentifrice — Each subject will use this product during one of the six treatment periods in the crossover study design.
  Arms: Colgate 1450 ppm Fluoride (1.1% sodium monofluorophosphate) Dentifrice
Drug: 1500 ppm MFP/CaCO3 1.16% sodium monofluorophosphate) Dentifrice — Each subject will use this product during one of the six treatment periods in the crossover study design.
  Arms: 1500 ppm MFP/CaCO3 1.16% sodium monofluorophosphate) Dentifrice
Drug: 1100 ppm (0.454% Stannous fluoride) Dentifrice — Each subject will use this product during one of the six treatment periods in the crossover study design.
  Arms: 1100 ppm (0.454% Stannous fluoride) Dentifrice

SUMMARY:
The primary objective is to compare the remineralization and demineralization inhibition potential of early subsurface carious lesions in enamel in situ after rinsing with six different aqueous slurries of toothpaste formulations.

ELIGIBILITY:
Inclusion Criteria:

* Be 18-75 years of age.
* Provide written informed consent prior to participation and be given a signed copy of the informed consent form.
* Be in good general health based on medical/dental history and oral exam.
* Have no history of adverse or allergic reactions to tin or tin-containing products.
* Agree not to participate in any other oral study for the study duration.
* Have a reasonable functional dentition as determined by the oral examiner and sufficient teeth to support the fabricated dental appliance.
* Be willing to participate in the study, able to follow the study directions, successfully tolerate/perform all study procedures, and willing to return for all specified visits at their appointed time.
* Be willing to refrain from using non-study dentifrice, mouth rinse, chewing gum, and other non-study oral care products during the study.
* Be willing to postpone all elective dental procedures until the study has been completed.
* Be willing to refrain from using calcium chews while using the test products.
* Be willing and able to refrain from wearing a nightguard (occlusal splint) for the entire course of the study (for nightguard wearers only).
* Ability to understand, and ability to read and sign, the informed consent form.
* Have at least 22 natural teeth.
* Have a gum-stimulated whole salivary flow rate ≥ 1.0 ml/minute and unstimulated whole salivary flow rate ≥ 0.2 ml/minute.

Exclusion Criteria:

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-07-31 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2023-12-11 (Actual)

PRIMARY OUTCOMES:
Mineral Density | 14 days
  The percent mineral profile of each enamel/dentinel slab's demineralized control and remineralized/treated lesion, obtained from the microdensitometry analysis, will be compared with the median sound enamel percent mineral profile of the same section. A negative value indicates mineral has been lost and, therefore, the lesion has progressed, whereas a positive value indicates mineral has been gained and, therefore, the lesion has regressed.
Scanning Electron Microscopy (SEM) | 14 days
  SEM imaging and SEM-EDS analysis will be conducted on TMR sections and whole sections of dentine lesions treated in situ to assess the occlusion of dentine tubules and distribution of elements within the lesions following the experiment.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Melbourne, Melbourne, Australia